CLINICAL TRIAL: NCT02116439
Title: Evaluation of the Manifestation of Patient Aggresivity in an Emergency Department
Acronym: ASAU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRIP/2013/MC-01; 1739572 v 0 (Other: CNIL number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Emergency Room
Keywords: Violence
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Violent events: People in this group were observed to manifest violence.
- Victims: People in this group are the victims of the other group.

SUMMARY:
The main objective of this study is to determine the average total number of violent events per observation period occurring in the emergency department at the Nîmes University Hospital. The list of violent events is pre-determined and based on a series of interviews with emergency department staff.

DETAILED DESCRIPTION:
This observational study will take place via a representative sample of 90 observation periods. One observation period consists of 7.5 consecutive hours between two team rotations during the day and 10 consecutive hours at night. These observational periods include the moment when health-care teams are debriefed during a shift-change, which we suspect to be a sensitive time point.

Observation periods are randomly selected over a period of 1 year, and stratified for time of day (morning, afternoon, evening), day of the week and month.

The secondary objectives of the observation phase are to identify factors associated with the average number of violent events per work period (number of patients attending the emergency department, time of staff debriefing during shift change, time of day, week or weekend, individual patient characteristics (gender, age, patient or accompanying a patient, waiting time from arrival in the emergency room to emergency consultation, reason for consultation), characteristics of victims of violence, characteristics of the health care team ...)

The anticipated total number of violent events is unknown at the beginning of the study; we indicated '50' as a guess.

ELIGIBILITY:
Inclusion Criteria:

* Persons manifesting violence according to a pre-determined list of watched-for events will be observed
* The victims of the above-mentioned violence will also be observed and interviewed

Exclusion Criteria:

* Persons not manifesting violence according to a pre-determined list of watched-for events

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons manifesting violence (and their victims) according to a pre-determined list of watched-for events will be observed.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2014-04-02 (Actual); Study Completion 2014-04-02 (Actual)

PRIMARY OUTCOMES:
The number of violent events occuring per work period | Baseline to end of period (maximum of 10 hours)

SECONDARY OUTCOMES:
Date | Baseline (hour 0)
Day of the week | Baseline (hour 0)
Time at the beginning of the observation period | Baseline (hour 0)
Number of male nurses present in the department | Baseline to end of observation period (maximum 10 hours)
Number of female nurses present in the department | Baseline to end of observation period (maximum 10 hours)
Number of nursing assistants present in the department | Baseline to end of observation period (maximum 10 hours)
Number of doctors present in the department | Baseline to end of observation period (maximum 10 hours)
Number of patients present in the department | Baseline (hour 0)
Number of accompaning persons (bringing in patients) present in the department | Baseline (hour 0)
Number of accompaning persons (bringing in patients) present in the waiting room | Baseline (hour 0)
Number of patients present in the department | End of observation period (maximum 10 hours)
Number of accompaning persons (bringing in patients) present in the department | End of observation period (maximum 10 hours)
Number of accompaning persons (bringing in patients) present in the waiting room | End of observation period (maximum 10 hours)
Time of day at the beginning of a staff debriefing during a shift change. | During an observation period (maximum 10 hours)
Time of day at the end of a staff debriefing during a shift change. | During an observation period (maximum 10 hours)
Time at the beginning of a violent event | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Time at the end of a violent event | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Was the event correctly declared according to current procedures? yes/no | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Sex (m/f) | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Is the person a patient or a person accompanying a patient? | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Reason why the patient is coming to the emergency department. | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Time (delay) patient has been waiting before manifestation of violence. | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.
Age (years) | During an observation period (maximum 10 hours)
  To be recorded for each event for each victim of a person manifesting violence.
Sex (m/f) | During an observation period (maximum 10 hours)
  To be recorded for each event for each victim of a person manifesting violence.
Years of work experience | During an observation period (maximum 10 hours)
  To be recorded for each event for each victim of a person manifesting violence.
Professional category | During an observation period (maximum 10 hours)
  To be recorded for each event for each victim of a person manifesting violence.
Presence/absence of difference in what was observed and what the victim remembers | 72 hours after a violent event
Violence severity scale | During an observation period (maximum 10 hours)
  To be recorded for each event for each person manifesting violence.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Chazel, Principal Investigator — CHRU de Nîmes - Hôpital Universitaire Carémeau
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Chazel M, Alonso S, Price J, Kabani S, Demattei C, Fabbro-Peray P. Violence against nurses in the emergency department: an observational study. BMJ Open. 2023 Apr 4;13(4):e067354. doi: 10.1136/bmjopen-2022-067354. PMID 37015789